CLINICAL TRIAL: NCT05032326
Title: Long-term Interventional Follow-up Study up to 4 Years of Age of Children With Prader-Willi Syndrome Included in the OTBB3 Clinical Trial and Comparison With an Untreated Cohort of Children With Prader-Willi Syndrome
Brief Title: Long-term Interventional Follow-up Study of Children With Prader-Willi Syndrome Included in the OTBB3 Clinical Trial
Acronym: OTBB3-FU
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0421
Record Dates: First submitted 2021-06-24; First posted 2021-09-02 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; Oxytocin
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OXYTOCIN (OT) Treated cohort (Other): babies treated with Oxytocin during the OTBB3 study
  Interventions: Drug: Follow-up study of the treated cohort
- Untreated cohort (Other): babies not included in the OTBB3 study and therefore never treated with Oxytocin
  Interventions: Other: Follow-up study of the untreated cohort

INTERVENTIONS:
Drug: Follow-up study of the treated cohort — follow-up study of the patients in the treated cohort: that have been included in the otbb3 study
  Arms: OXYTOCIN (OT) Treated cohort
Other: Follow-up study of the untreated cohort — follow-up study of the patients in the untreated cohort: that have NOT been included in the otbb3 study
  Arms: Untreated cohort

SUMMARY:
This study is a prospective, multicentre, interventional cohort study in children with Prader-Willi Syndrome (PWS) over 4 years (no treatment administered). The duration of the preceding OTTB3 study is 26 weeks. An untreated cohort of children with PWS will be included at an age of 2 years and followed up until an age of 4 years.

Regarding the untreated cohort, children with PWS born in France and too old to be recruited in OTBB3 trial, principally those who were born within one year before the start of OTBB3 trial, will be offered to participate in this study. Infants born later who couldn't be included in OTBB3 study will be also offered to participate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female child with a genetically confirmed diagnosis of PWS (patients can be enrolled if the genetic subtype is not available at inclusion, but the genetic subtype needs to be confirmed during the study);
2. The parents (or legal representative) must have signed the consent form;
3. Treated cohort: the child participated in the OTBB3 study and is aged 16±4 months at inclusion,
4. Untreated cohort: the child has never received OT, is aged 30±6 months at inclusion (in order to maximise the number of children in the untreated cohort) and is followed in France.

Exclusion Criteria:

1. Administrative problems:

   1. Inability for the parents (or legal representative) to understand/fulfil study requirements;
   2. No coverage by a social security regime;
2. Refusal of parents (or legal representative) to sign the consent form;

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2021-09-07 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Confirmation of the long term safety profile (1) | 4 years
  The number of patients with adverse events (AEs)
Confirmation of the long term safety profile (2) | 4 years
  The percentage of patients with adverse events (AEs)
Confirmation of the long term safety profile (3) | 4 years
  Assessment in the treated cohort of the occurrence of the main comorbidities in Prader Willi Syndrome
Confirmation of the long term safety profile (4) | 4 years
  Assessment in the treated cohort of:
  The occurrence of medications, surgery and rehabilitations by collecting type, age (years) at start and stop, dosing or frequency

SECONDARY OUTCOMES:
Complete the safety assessment by the description of the development of the child (1.1) | 4 years
  Assessment in the treated cohort of: weight (kilograms)
Complete the safety assessment by the description of the development of the child (1.2) | 4 years
  Assessment in the treated cohort of: height (meters)
Complete the safety assessment by the description of the development of the child (1.3) | 4 years
  Assessment in the treated cohort of: BMI (kg/m^2)
Complete the safety assessment by the description of the development of the child (2.1) | 4 years
  Assessment in the treated cohort of Child development: age at which sitting has been reached
Complete the safety assessment by the description of the development of the child (2.2) | 4 years
  Assessment in the treated cohort of Child development: age at which crawling has been reached
Complete the safety assessment by the description of the development of the child (2.3) | 4 years
  Assessment in the treated cohort of Child development: age at which walking has been reached
Complete the safety assessment by the description of the development of the child (2.4) | 4 years
  Assessment in the treated cohort of Child development: age at which running has been reached
Complete the safety assessment by the description of the severity of the disease | 4 years
  Severity of the disease for:
  Eating disorders by using Hyperphagia Questionnaire for Clinical Trials (HQCT);
Complete the safety assessment by the description of the severity of the disease (2) | 4 years
  Severity of the disease for:
  Psychiatric disorders by using the Child Behaviour Checklist (CBCL);
Assessment of endocrine disorders by IGF1 | 4 years
  Analysis of plasma Insulin-like growth factor 1 (IGF1, ng/mL)
Assessment of endocrine disorders by TSH | 4 years
  Analysis of plasma thyroid stimulating hormone (TSH, µUI/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Maithé TAUBER, MD, Principal Investigator — University Hospital, Toulouse
Locations (12):
- France (12):
  - Hôpital Femme Mère Enfant, Bron
  - CHU Dijon Hôpital des Enfants, Dijon
  - CHU de Grenoble, Grenoble
  - Hôpital Jeanne de Flandre, Lille
  - Hôpital de la Timone Enfant, Marseille
  - CHU Nancy, Nancy
  - CHU Nantes, Nantes
  - Hôpital CHU-Lenval, Nice
  - Groupe Hospitalier Necker - Enfants Malades, Paris
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - Centre de réfrence Prader-Willi, Hospital of infants, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided